CLINICAL TRIAL: NCT06155890
Title: Restoring Mobility: Roles of Percutaneous Consolidation for Pelvic Ring Bone Lesions -a Multicenter Study
Brief Title: Restoring Mobility: Roles of Percutaneous Consolidation for Pelvic Ring Bone Lesions
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 23Imagerie02
Record Dates: First submitted 2023-11-15; First posted 2023-12-05 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2023-11

CONDITIONS: Pelvic Ring Tumor Lesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate early functional outcomes following percutaneous screw fixation or cementoplasty for pelvic ring tumor lesions.

ELIGIBILITY:
Inclusion :

- Individuals with cancer who underwent percutaneous screw fixation or cementoplasty either for prophylactic consolidation or treatment of pathologic fractures in pelvic ring tumors.

Exclusion criteria :

* minors
* incompetent adults
* refused to participate in the study
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with cancer who underwent percutaneous screw fixation or cementoplasty either for prophylactic consolidation or treatment of pathologic fractures in pelvic ring tumors.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2023-09 (Actual); Study Completion 2023-10 (Actual)

PRIMARY OUTCOMES:
postoperative weight-bearing ambulation | During hospitalization, mainly less than 3 days
  the ability of the patient to walk and bear weight after the procedure and its associated timeframe.

SECONDARY OUTCOMES:
Adverse event | During hospitalization, and follow-up
  adverse event during procedure or hospitalization
Duration of hospitalization | Mainly less than 3 days
  The duration of hospitalization will be measured between the day and time of arrival at the hospital and the day and time of discharge from the hospital
Long-term effectiveness in preventing pathological fractures of the pelvic ring | 3 months after the procedure, and during follow-up, up to 5 years
  Absence of pelvic ring fracture during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- CHU NICE, Nice, France

REFERENCES:
- [Derived] Dien E, Stacoffe N, Pavan LJ, Torre F, Ranc PA, Vivarrat-Perrin T, Chalamet B, Pialat JB, Kastler A, Amoretti N. Restoring mobility: roles of percutaneous consolidation for pelvic ring bone lesions-a multicenter study. Eur Radiol. 2025 Jun;35(6):3270-3281. doi: 10.1007/s00330-024-11193-6. Epub 2024 Nov 21. PMID 39567430